CLINICAL TRIAL: NCT03257228
Title: The Association Between Diabetes Mellitus, Oral Lichen Planus and Insulin-like Growth Factors 1 and 2 (IGF1 and IGF2)
Status: Completed | Type: Observational
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Božana Lončar Brzak, Asisstant Professor, University of Zagreb
Other Study IDs: BM 1.62
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Oral Lichen Planus; Diabetes Mellitus
MeSH Terms: conditions — Lichen Planus, Oral; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsy samples of oral mucosa
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- oral lichen planus and diabetes mellitus: Histopathologically confirmed samples of oral lichen planus underwent immunohistochemical analysis of IGF1 and IGF2 expression. Blood glucose level was determined one day before taking biopsy.
  Interventions: Genetic: comparative semiquantitative immunohistochemistry
- oral lichen planus: Histopathologically confirmed samples of oral lichen planus underwent immunohistochemical analysis of IGF1 and IGF2 expression. Blood glucose level was determined one day before taking biopsy.
  Interventions: Genetic: comparative semiquantitative immunohistochemistry
- healthy mucosa: Samples of healthy mucosa underwent immunohistochemical analysis of IGF1 and IGF2 expression. Blood glucose level was determined one day before taking mucosa samples.
  Interventions: Genetic: comparative semiquantitative immunohistochemistry

INTERVENTIONS:
Genetic: comparative semiquantitative immunohistochemistry

SUMMARY:
Diabetes mellitus is among the most common chronic diseases, with significant and well documented impact on oral cavity health. Among the most common diseases of the oral cavity mucosa and complications in patients with impaired glucose metabolism and diabetes mellitus is oral lichen ruber (OLR), which according to World Health Organisation (WHO) is considered potentially malignant disorder. It was found that lichen ruber in diabetes mellitus has a much more aggressive clinical course in the form of atrophic-erosive and ulcerative lesions showing an increased tendency to malignant transformation. Although OLR etiology is unknown, evidence suggests cell-mediated autoimmune pathogenesis. OLR epithelial cells show anomalies in both enzymatic activity and carbohydrate metabolism, which may be related to hormones regulating carbohydrate, insulin and insulin-like growth factors 1 and 2 (IGF-1 and IGF-2) metabolism. The hypothesis of our research is that patients with diabetes mellitus and oral lichen ruber lesions will have a disturbance of insulin-like growth factors 1 and 2 and hence a greater risk of malignant transformation, compared to patients with oral lichen ruber without diabetes and healthy patients without alterations in the oral mucosa.

DETAILED DESCRIPTION:
Oral lichen ruber (OLR) in the diabetes mellitus patients has more aggressive clinical course in the form of atrophic-erosive and ulcerative lesions showing an increased tendency to malignant transformation. OLR epithelial cells show anomalies in both enzymatic activity and carbohydrate metabolism, which may be related to hormones regulating carbohydrate, insulin and insulin-like Growth Factors 1 and 2 (IGF-1 and IGF-2) metabolism. The role of insulin-like growth factors (IGFs) is of great importance in normal growth and cell development (cell proliferation, differentiation and apoptosis), and is involved in different aspects of cell transformation in malignant phenotype. A change in the expression of IGF1, IGF2 and IGF2R proteins is described in several types of malignant tumors including oral cancer. However, data on their role in the development of malignant lesions of the oral cavity are scarce, and the results are inconsistent. Our hypothesis is that patients with diabetes mellitus and oral lichen ruber lesions will have a disturbance of insulin-like growth factors 1 and 2 and hence a greater risk of malignant transformation, compared to patients with oral lichen ruber without diabetes and healthy patients without alterations in the oral mucosa.

ELIGIBILITY:
Inclusion Criteria:

* histopathologically confirmed oral lichen ruber patients, with and without diabetes mellitus
* healthy volunteers referred for alveolotomy

Exclusion Criteria:

* non-consent patients

Ages: 30 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients included in the study are patients with oral lichen ruber referred to the Department of Oral Medicine, University of Zagreb. Healthy mucosa samples were taken from healthy volunteers referred for alveotomy of wisdom tooth to the Department of Oral Surgery, School of Dental Medicine, University of Zagreb.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2015-11-01 (Actual); Study Completion 2015-11-01 (Actual)

PRIMARY OUTCOMES:
Insulin like growth factors in patients with OLP and diabetes mellitus | 2014-2015
  Evaluation of the Insulin-like growth factor 1 and 2 (IGF1 and IGF 2) in patients with oral lichen planus and diabetes mellitus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Djiogue S, Nwabo Kamdje AH, Vecchio L, Kipanyula MJ, Farahna M, Aldebasi Y, Seke Etet PF. Insulin resistance and cancer: the role of insulin and IGFs. Endocr Relat Cancer. 2013 Jan 7;20(1):R1-R17. doi: 10.1530/ERC-12-0324. Print 2013 Feb. PMID 23207292
- [Background] Cohen DH, LeRoith D. Obesity, type 2 diabetes, and cancer: the insulin and IGF connection. Endocr Relat Cancer. 2012 Sep 5;19(5):F27-45. doi: 10.1530/ERC-11-0374. Print 2012 Oct. PMID 22593429
- [Background] Sarfstein R, Friedman Y, Attias-Geva Z, Fishman A, Bruchim I, Werner H. Metformin downregulates the insulin/IGF-I signaling pathway and inhibits different uterine serous carcinoma (USC) cells proliferation and migration in p53-dependent or -independent manners. PLoS One. 2013 Apr 19;8(4):e61537. doi: 10.1371/journal.pone.0061537. Print 2013. PMID 23620761